CLINICAL TRIAL: NCT03938285
Title: Effect of Hemodiafiltration Plus MCOs on Uremic Toxins Rem
Brief Title: Effect of Hemodiafiltration Plus MCOs on Uremic Toxins Removal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Collaborators: Renal Research Institute (Other)
Responsible Party: Principal Investigator, Magdalena Madero, Head of Nephrology, Instituto Nacional de Cardiologia Ignacio Chavez
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PT-19-103
Record Dates: First submitted 2019-05-02; First posted 2019-05-06 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Hemodiafiltration; Chronic Kidney Disease Requiring Chronic Dialysis

STUDY DESIGN:
Intervention Model Description: 12 patients will be included, they will be divided in 4 groups: high flux HD, extended HD (HDx), OL-HDF, and OL-HDF with medium cut-off membrane. All sessions will be performed in a 5008S CorDiax that enables HD and OL-HDF, we will use an FX CorDiax 80 dializer (effective area 1.8 m2) for OL-HDF and conventional HD, and the Theranova 400 dializer (effective area 1.7 m2)for OL-HDF with medium cut-off membrane, and HDx. Every patient will be in each of the 4 groups, and they will receive 3 sessions in each group. Every session will have a duration of 240 minutes with a Qb of 300 mL/min. Blood samples will be drawn in every session, every blood sample will consist of 4-6 mL of EDTA plasma; this volumen would include 0.5 mL for biobanking, blood will be drawn from the arterial, and venous outlet, and a dialysate sample will be drawn in every time point.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- High Flux Hemodialysis (Active Comparator): High Flux Hemodialysis with an FxCordiax 120 membrane, with Qb of 350, 4 hours of treatment.
  Interventions: Other: FxCordiax 120 membrane
- Extended Hemodialysis (Active Comparator): Extended Hemodialysis with a Theranova 400 membrane, with Qb of 350, 4 hours of treatment.
  Interventions: Other: Theranova 400 membrane
- On Line Hemodiafiltration (Active Comparator): On Line Hemodiafiltration with an FxCordiax 120 membrane, with Qb of 350, 4 hours of treatment, and post filter substitution rate of 20-21 liters.
  Interventions: Other: FxCordiax 120 membrane
- On Line Hemodiafiltration with an MCO membrane (Active Comparator): On Line Hemodiafiltration with a Theranova 400 membrane, with Qb of 350, 4 hours of treatment, and post filter substitution rate of 20-21 liters.
  Interventions: Other: Theranova 400 membrane

INTERVENTIONS:
Other: Theranova 400 membrane — Patients will receive 4 different dialysis treatment, HD with a high flux membrane, extended HD, On Line Hemodiafiltration, and the novel On Line Hemodiafiltration with an MCO membrane.
  Arms: Extended Hemodialysis; On Line Hemodiafiltration with an MCO membrane
Other: FxCordiax 120 membrane — Patients will receive 4 different dialysis treatment, HD with a high flux membrane, extended HD, On Line Hemodiafiltration, and the novel On Line Hemodiafiltration with an MCO membrane.
  Arms: High Flux Hemodialysis; On Line Hemodiafiltration

SUMMARY:
Conventional hemodialysis is essential for the treatment of ESRD patients by reducing serum concentration of uremic toxins and correcting fluid overload. Nevertheless, HD removes almost exclusively low-range uremic toxins. Convective methods might reduce complications associated to molecules of medium-range molecular weight. On-Line Hemodiafiltration (OL-HDF) is the result of the combination between convection and diffusion, this modality allows better clearence of middle-range molecules, and protein bound molecules with better hemodynamic tolerance, but at higher cost. In order to solve this problem the middle cut-off membranes were developed, achieving cleareance of molecules between 15,000 to 40,000 Da with low albumin loss. To our knowledge no study has ever evaluated the use of middle cut-off membranes on OL-HDF. This is a prospective, experimental study which will include 12 patients with ESRD that receive OL-HDF treatment on the National Institute of Cardiology "Ignacio Chavez" OL-HDF Unit. They will be divided in 4 groups: high flux HD, extended HD (HDx), OL-HDF, and OL-HDF with medium cut-off membrane.

DETAILED DESCRIPTION:
Introduction:

The Kidney Disease Improved Global Outcomes (KDIGO) defines Chronic Kidney Disease (CKD), as a decline of the glomerular filtration rate (GFR) below 60 mL/min/1.72 m2SC, associated with structural or functional abnormalities in a period greater than three months. CKD it's classified in 5 stages based con GFR and albuminuria . Stage 5 is considered the end stage, and it's also known as End Stage Renal Disease (ESRD), in this stage usually the patients require some kind of renal function replacement (RFR), otherwise CKD will cause the death of the patient.

In Mexico the principal cause of CKD is Type 2 Diabetes Mellitus (DM2), closely followed by Systemic Arterial Hypertension (SAH), according to the 2012 National Survey of Health and Nutrition (ENSANUT) from Mexico there are 6.4 million adults with DM2, and 22.4 million adults with SAH. In Mexico the prevalence of patients currently receiving RFR it's unknown, but based in different sources we estimate that 129 thousand patients have ESRD, and only 60 thousand receive some kind of RFR therapy.

In Mexico (based on data published by the Mexican Institute of Social Security), 41% of the dialysis patients are on hemodialysis (HD). ESRD patients on HD have a greater incidence of cardiovascular outcomes which cause an important impact on survival. This increase on cardiovascular outcomes can be explained by the high prevalence in this population of type 2 diabetes mellitus, and hypertension, as well as adverse outcomes associated with uremia such as chronic inflammation, and bone mineral disease vascular calcifications.

Uremic toxins are clasiffied according to their molecular weight in low-range molecules (< 500 Da), middle-range molecules (500 Da - 60 kDa), hydrosoluble molecules, and protein bound molecules.

Conventional hemodialysis is essential for the treatment of ESRD patients by reducing serum concentration of uremic toxins and correcting fluid overload. Nevertheless, HD removes almost exclusively low-range uremic toxins. Convective methods might reduce complications associated to molecules of medium-range molecular weight.

On-Line Hemodiafiltration (OL-HDF) is the result of the combination between convection and diffusion, this modality allows better clearence of middle-range molecules, and protein bound molecules with better hemodinamic tolerance. The ES-HOL study showed that OL-HDF with post-filter sustitution patients had lower mortality in comparision with conventional HD.

Convection can be poorly efficient when there´s disturbances on blood flow, time of dialysis, and low dialyser quality, to solve this kind of issues newer dialysers with better cut-offs had been developed, with this new dialysers one can achieve better clearence and greater sustitution volumes. This new dialysers allow clearence of middle-range and protein bound molecules like inflamatory mediators in sepsis, and light weigth chain immunoglobulins. Nevertheless this new dialysers cause high protein loss.

In order to solve this problem the middle cut-off membranes were developed, achieving cleareance of molecules between 15,000 to 40,000 Da with low albumin loss.

Recently our knowledge on uremic toxins has grown importantly, this increase in knowledge is due in part to the creation of international collaboration groups such as the European Uremic Toxin Work Group (EuTOX), which has recently described over 130 uremic toxins. Also urea metabolomics had made important contributions describing the metabolism of uremic toxins in plasma. One study used metabolomics to evaluated over 80 HD sessions, showing an important description of the metabolism of uremic toxins.

To our knowledge no study has ever evaluated the use of middle cut-off membranes on OL-HDF. This study aimes to show that the combination of OL-HDF with middle cut-off membranes can achieve a higher cleareance of middle-bound molecules in comparison to regular OL-HDF with out affecting the nutritional status of the patients.

Study design This is a prospective, experimental study which will include 12 patients with ESRD that receive OL-HDF treatment on the National Institute of Cardiology "Ignacio Chavez" OL-HDF Unit.

Inclusion Criteria:

* Age greater or equal to 18 years.
* Patients that receive OL-HDF three times per week.
* Patients with no residual uresis.
* Hemoglobin greater that 7 g/L.
* Patients that can exercise during treatment.
* Patients must sign informed consent.

Exclusion Criteria:

* Age less tan 18.
* Presence of residual uresis.
* Hb less that 7 g/L.
* Patients incapable of exercising during dialysis.

Elimination Criteria:

* Hospitalization of any cause during the study.
* Patients incapable of finishing a dialysis session.

Methods:

12 patients will be included, they will be divided in 4 groups: high flux HD, extended HD (HDx), OL-HDF, and OL-HDF with medium cut-off membrane. All sessions will be performed in a 5008S CorDiax that enables HD and OL-HDF, we will use an FX CorDiax 80 dializer (effective area 1.8 m2) for OL-HDF and conventional HD, and the Theranova 400 dializer (effective area 1.7 m2)for OL-HDF with medium cut-off membrane, and HDx. Every patient will be in each of the 4 groups, and they will receive 3 sessions in each group. Every session will have a duration of 240 minutes with a Qb of 300 mL/min. Blood samples will be drawn in every session at the following time points 5, 30, 60, 120 180, and 240 minutes, every blood sample will consist of 4-6 mL of EDTA plasma; this volumen would include 0.5 mL for biobanking, blood will be drawn from the arterial, and venous outlet, and a dialysate sample will be drawn in every time point.

Samples will we packed, refrigerated and send to the Renal Research institute Lab, for uremic toxins metabolomics analysis, as well as middle-range uremic molecules, such as Beta 2 mycroglobulin, albumin, vitamin B12, myoglobin, Cystatin C, Urea Nitrogen, and Uric Acid.

Every patient will have a full nutritional assesment before the first session, and after the third session of every modality; the assesment will include electric bioimpedance for determination of ECW/TBW, and phase angle, dinamometry, nutritional plan, and MIS (Malnutrition Inflammation Score) score.

Statistical Analysis:

For statistical analysis we will use the software STATA 13.0. Quantitative variables will be analized with Shapiro-Wilk, Student T will be used for group comparations. We will consider a p value of significance of less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age greater or equal to 18 years.
* Patients that receive OL-HDF three times per week.
* Patients with no residual uresis.
* Hemoglobin greater that 7 g/L.
* Patients that can exercise during treatment.
* Patients must sign informed consent.

Exclusion Criteria:

* Age less tan 18.
* Presence of residual uresis.
* Hb less that 7 g/L.
* Patients incapable of exercising during dialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Uremic Toxins Clearance | 1 month
  The combination of On Line Hemodiafiltration with an MCO membrane will have a better sieving coefficient for middle and protein bound molecules in comparison with other dialysis modalities.

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Madero, MD, Principal Investigator — Instituto Nacional de Cardiologia
Locations (2):
- Mexico (2):
  - Instituto Nacional de Cardiologia Ignacio Chávez, Mexico City
  - Instituto Nacional de Cardiología Ignacio Chávez, México

IPD SHARING:
Plan to Share IPD: Undecided
We haven´t decided what information will be disclosed on advance.

REFERENCES:
- [Derived] Armenta-Alvarez A, Lopez-Gil S, Osuna I, Grobe N, Tao X, Ferreira Dias G, Wang X, Chao J, Raimann JG, Thijssen S, Perez-Grovas H, Canaud B, Kotanko P, Madero M. Removal of Middle Molecules and Dialytic Albumin Loss: A Cross-over Study of Medium Cutoff and High-Flux Membranes with Hemodialysis and Hemodiafiltration. Kidney360. 2023 Aug 1;4(8):1095-1102. doi: 10.34067/KID.0000000000000185. Epub 2023 Jun 12. PMID 37651666